CLINICAL TRIAL: NCT02200562
Title: A Phase I/II Study of Concurrent Ipilimumab and Dabrafenib in Unresectable Stage III or Stage IV Melanoma
Brief Title: Ipilimumab and Dabrafenib in the 1st Line Tx of Unresectable Stage III/IV Melanoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: BMS withdrew support and required this trial to stop enrolling; Phase II portion never began, only a Phase I trial.
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI68132
Record Dates: First submitted 2014-03-27; First posted 2014-07-25 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Stage III or IV Melanoma
MeSH Terms: interventions — Ipilimumab; dabrafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ipilimumab and Dabrafenib (Experimental)
  Interventions: Drug: ipilimumab and dabrafenib

INTERVENTIONS:
Drug: ipilimumab and dabrafenib

SUMMARY:
Phase I/II study of ipilimumab concurrent ipilimumab and dabrafenib as first line treatment in Stage III or IV melanoma.

Assessing safety of Ipilimumab and dabrafenib in combination. Also, assessing disease control rates.

ELIGIBILITY:
Inclusion Criteria:

* For Phase I: Locally advanced or metastatic BRAF V600E/K/R positive melanoma that is either treatment-naïve or treatment-experienced. For the latter, progression, or stable as best response, or intolerance to the last treatment is required. Previous treatments can be local or systemic therapies. There are no limits to the number of prior therapies. For all patients, disease does not have to be measurable but must be evaluable, which is defined as one or more lesions which are known to be present, but which cannot be measured. eg: Bony lesions, pleural effusion, ascites.
* For Phase I: For treatment-experienced patients, the following washout periods are required prior to enrollment on the study: 2 weeks wash out after prior local therapy (such as radiation therapy or intra-lesional therapy), 4 weeks wash out after cytotoxic therapy or high dose interleukin-2, and 6 weeks wash out after anti-PD-1 or anti-PD-L1 therapy. For all other therapy not mentioned, a wash out period of at least 5 half lives will be needed.
* For phase II: Histological diagnosis of BRAF V600E/K melanoma, unresectable stage III or stage IV, according to the AJCC Staging Manual, 7th Edition, 2011. Must have measurable disease, and no prior systemic treatment for locally advanced or metastatic melanoma. Previous local therapy is allowed. Previous systemic treatment for any stage III disease that was subsequently rendered NED (no evidence of disease) by surgery is allowed except for ipilimumab and BRAF inhibitors. Patients with resectable disease who do not want surgery for any reason are also allowed. Measurable disease is defined as least one lesion that can be accurately measured in two dimensions with both diameters greater than 1.0cm. For CT/MRI evaluations, an effective slice thickness is required of less than or equal to 5 mm. For slice thickness greater than 5mm, both diameters must be greater than or equal to 2.0cm at baseline.
* ECOG performance status 0, 1 or 2
* Negative pregnancy test for women of childbearing potential within 7 days of starting study treatment.
* Lab testing results in accordance with protocol WBC greater/equal to 2,000/mm3 ANC greater/equal to 1200/mm3 Platelet greater/equal 1000,000/mm2 Hemoglobin greater/equal 9 gm/dL (may be transfused) Serum bilirubin levels less/equal 1.5 mg/dL except for patients with Gilbert's syndrome.
* Serum aspartate transaminase (AST) and serum alanine transaminase (ALT) less/equal 2.5 X upper limit of normal Alkaline phosphatase less/equal 2.5 times upper limit of normal Serum Creatinine levels less/equal 1.5 mg/dL Left Ventricular Ejection Fraction (LVEF) greater or equal to lower limit of normal by ECHO Women of childbearing potential should be advised to avoid becoming pregnant and men should be advised to not father a child while receiving treatment with ipilimumab or dabrafenib. Patients should agree to use an appropriate method of birth control while on study.
* Age greater than 18 years and of any gender or race. Able to provide informed consent and have signed an approved consent form that conforms to federal and institutional guidelines.

Exclusion Criteria:

* Concurrent therapy with any other non-protocol anti-cancer therapy
* Prior systemic treatments with either ipilimumab or a BRAF inhibitor (such as vemurafenib or dabrafenib).
* Prior local therapy within 2 weeks (for both phases I and II) or prior systemic therapy within 4 weeks of starting protocol treatment (phase I).
* For phase II: Any prior systemic therapy for locally advanced or metastatic melanoma. Prior local therapy such as radiation or intratumoral injection is allowed. Previous systemic treatment for any stage III disease that was subsequently rendered NED (no evidence of disease) by surgery is allowed.
* Brain metastases (except if all known lesions were previously treated with surgery or stereotactic radiosurgery and lesions, if still present, are confirmed stable for greater than or equal to 2 weeks prior to enrollment, and are asymptomatic with no corticosteroid requirements for greater than or equal to weeks prior to randomization, and no enzyme inducing anticonvulsants for greater than or equal to 2 weeks prior to randomization). Brain MRI or CT is required at screening.
* Anyone with a second malignancy expected to require cytotoxic chemotherapy or immune modulating therapy within 3 months of enrollment
* Pre-existing autoimmunity: History of inflammatory bowel disease; history of symptomatic autoimmune disease (e.g., rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, autoimmune vasculitis [e.g., Wegener's Granulomatosis]); motor neuropathy considered of autoimmune origin (e.g., Guillain-Barre Syndrome). Subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
* No concurrent systemic corticosteroids (or other systemic immunosuppressant's), including oral steroids (i.e. prednisone, dexamethasone), continuous use of topical steroid creams or ointments, or ophthalmologic steroids. If a subject is currently taking corticosteroids, treatment should be discontinued two weeks prior to starting protocol therapy. Occasional use of steroid inhalers is allowed.
* Any serious or uncontrolled medical disorder or active infection that, in the opinion of the investigator, may increase the risk associated with study participation, study drug administration, or would impair the ability of the subject to receive protocol therapy.
* Any known positive test for hepatitis B virus or hepatitis C virus indicating acute or chronic infection. Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
* Herbal remedies (e.g., St. John's wort) within 1 week of enrollment.
* Drugs that are strong inhibitors or inducers of CYP3A or CYP2C8, p-glycoprotein (Pgp) or Bcrp transporter because they may alter dabrafenib concentrations. The list may be modified based on emerging data; consider therapeutic substitutions for these medications. Patients must be off treatment for at least 1 week prior to enrollment.
* A history of known glucose-6-phosphate dehydrogenase (G6PD) deficiency.
* The presence of any other medical or psychiatric disorder that, in the opinion of the treating physician, would contraindicate the use of the drugs in this protocol or place the subject at undue risk for treatment complications
* Pregnancy or breast feeding
* A history of a severe hypersensitivity reaction to ipilimumab or dabrafenib
* Any reason why, in the opinion of the investigator, the patient should not participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-12; Primary Completion 2017-01-20 (Actual); Study Completion 2017-01-20 (Actual)

PRIMARY OUTCOMES:
Safety of ipilimumab and dabrafenib in combination | Safety analysis will be measured based on frequency and severity of adverse events experienced by patients during the study treatment period which is expected to last about 24 weeks.
  All patients who receive any study treatment will be included in the final summaries and listings of safety data. Detailed information collected for each AE will include a description of the event, duration, severity, relatedness to study drugs, action taken, and clinical outcome. Severity of the AEs will be graded according to the CTCAE version 4.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States